CLINICAL TRIAL: NCT04943354
Title: Associations of Combinations of Single-nucleotide Polymorphisms and Behavioural Risk Factors With Non-communicable Diseases and Adverse Outcomes in Women With Premature Ovarian Failure
Brief Title: Associations of Combinations of Single-nucleotide Polymorphisms in Women With Premature Ovarian Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 20-315-90017
Record Dates: First submitted 2020-11-27; First posted 2021-06-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2022-07

CONDITIONS: Primary Ovarian Insufficiency; Cardiovascular Diseases; Menopause, Premature; Coronary Disease; Pulmonary Embolism; Arrhythmias, Cardiac; Polymorphism, Single Nucleotide
Keywords: premature ovarian failure; hypoestrogenism; artificial menopause; cardiovascular disease; chronic non-infectious disease; cardiovascular outcomes; coronary heart disease; pulmonary embolism; cardiac arrhythmias; heart rhythm disturbances; single nucleotide polymorphisms
MeSH Terms: conditions — Primary Ovarian Insufficiency; Cardiovascular Diseases; Menopause, Premature; Coronary Disease; Pulmonary Embolism; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Women diagnosed with premature ovarian failure were selected from different medical institutions in Ryazan and the Ryazan region, all information was communicated to them in a clear and understandable way and they also signed an informed voluntary consent. Premature ovarian failure - defined as the occurrence of secondary amenorrhoea ≥4 months at the age of under 45 years together with FSH levels above 40 IU/L.
  Inclusion criteria were: female gender, age at menopause < 45 years, onset of secondary amenorrhoea ≥ 4 months, FSH levels higher than 40 IU/l, or a previous diagnosis of premature ovarian failure.
  The control group was formed based on comparability criteria of gender, age and BMI to minimise the influence of phenotype on the results. The control group consisted of women without signs of PEN, so we aimed to compare the health status of these two different groups of women.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study of single-nucleotide polymorphisms in women diagnosed with premature ovarian failure (Active Comparator): Study of genes affecting single nucleotide polymorphisms: Reninangiotensin-aldosterone system (AGT, ACE), endothelial dysfunction (NOS3, EDN1), thrombosis-associated (ITGB3, ITGA2, FGB, GPIBA, SERPINE PAI1), proinflammatory (CRP, IL17A, IL2, IL10 1, IL10 2, TNFα, CRP 4, IL6, TLR2, TLR3, TLR4, TLR6, TLR9) in the study group of women diagnosed with premature ovarian failure.
  Interventions: Behavioral: Taking a person's venous blood
- Study of single-nucleotide polymorphisms in a control group of healthy women (Active Comparator): Study of genes affecting single nucleotide polymorphisms: Reninangiotensin-aldosterone system (AGT, ACE), endothelial dysfunction (NOS3, EDN1), thrombosis-associated (ITGB3, ITGA2, FGB, GPIBA, SERPINE PAI1), pro-inflammatory (CRP, IL17A, IL2, IL10 1, IL10 2, TNFα, CRP 4, IL6, TLR2, TLR3, TLR4, TLR6, TLR9) in a control group of healthy women .
  Interventions: Behavioral: Taking a person's venous blood

INTERVENTIONS:
Behavioral: Taking a person's venous blood — Collection of 5 ml of the patient's venous blood, carried out according to standard rules.

SUMMARY:
Research objective.

- To study the associations between combinations of single nucleotide polymorphisms and behavioural risk factors with non-communicable diseases and adverse outcomes in women with premature ovarian failure.

Research objectives:

* To study the associations between combinations of single-nucleotide polymorphisms and behavioural risk factors with heart rate disorders and adverse outcomes in women with premature ovarian failure
* Examine the associations between combinations of single nucleotide polymorphisms and behavioural risk factors with stable STIs in women with premature ovarian failure.
* Examine the associations between combinations of single nucleotide polymorphisms and behavioural risk factors with thrombomolia in women with premature ovarian failure
* Study the associations between combinations of single nucleotide polymorphisms and behavioural risk factors and adverse cardiovascular outcomes in women with premature ovarian failure.

DETAILED DESCRIPTION:
Methods of research:

* Questionnaire .
* Clinical examination
* Blood levels of sex hormones
* Blood lipid spectrum
* Coagulogram
* Glycemic profile
* EchoCG
* SMAD
* ECG
* Daily ECG monitoring
* Questionnaire EQ-5D
* Single-nucleotide polymorphisms of genes of the reninangyotensin-aldosterone system group (AGT, ACE), endothelial dysfunction (NOS3, EDN1), thrombosis-associated (ITGB3, ITGA2, FGB, GPIBA, SERPINE PAI1), pro-inflammatory (CRP, IL17A, IL2, IL10 1, IL10 2, TNFα, CRP 4, IL6, TLR2, TLR3, TLR4, TLR6, TLR9) polymorphisms.

Subject of study.

Women under 45 with Premature Ovarian Failure (PED). It is planned to include 615 people in the study. The study will have both prospective and retrospective parts. Patients will be divided into 4 groups:

* Women with OED without cardiovascular disease
* Women with OAI who have cardiovascular disease
* Control group No 1 Women with normal ovarian function without cardiovascular disease.
* Control group 2 Women with normal ovarian function without cardiovascular disease.

The groups will be comparable in number. All data obtained will be calculated for each group separately. A comparative analysis will then be made for all four groups.

Traditional risk factors, existing non-communicable diseases and the quality of life of patients will be identified using standard research methods.

The selected polymorphism groups are associated with various pathological processes leading to unfavourable cardiovascular outcomes. Their role has not been assessed in patients with premature ovarian failure.

The power of the study was calculated based on the expected number of adverse outcomes.

The division of patients into groups is related to the need to compare and evaluate unfavourable outcomes and non-communicable diseases in patients in order to create a risk scale.

ELIGIBILITY:
Inclusion Criteria:

* women under 45 years old
* presence of premature ovarian insufficiency in the medical history

Exclusion Criteria:

* male gender
* age over 45 years

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 238 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Age (years) | 2 year
  Patient age in years

SECONDARY OUTCOMES:
Menarche (years) | 2 year
  Age of onset of menarche expressed in years

OTHER OUTCOMES:
Pregnancy (number) | 2 year
  Number of pregnancies in history
Childbirth (number) | 2 year
  Number of pregnancies that ended in childbirth
Menopause (yes/no) | 2 year
  Current presence or absence of menopause
Surgical removal of both ovaries (yes/no) | 2 year
  History of surgery involving bilateral removal of both ovaries
Presence of amenorrhoea (at least 4 months) (yes/no) | 2 year
  A history of amenorrhoea for at least 4 months
Follicle stimulating hormone (FSH) level (mMed/ml) | 2 year
  Blood follicle-stimulating hormone content expressed in mMED/ml
Age at menopause (years) | 2 year
  Age of onset of menopause
Length of post-menopause (years) | 2 year
  How many years a person has been in the post-menopausal phase
Taking oral contraceptives (yes/no) | 2 year
  Whether the patient is continuously taking oral contraceptives
Taking hormone replacement therapy (HRT) (yes/no) | 2 year
  Whether the patient is taking regular hormone replacement therapy
Length of time on hormone replacement therapy (years) | 2 year
  How long the patient has been on hormone replacement therapy
Smoking status (yes/no) | 2 year
  Does the patient use nicotine-containing substances on a regular basis
Number of cigarettes smoked per day (number) | 2 year
  How many cigarettes the patient smokes per day on average
Smoking experience (years) | 2 year
  Number of years of active nicotine use by the patient
Smoking index (points) | 2 year
  Calculated as the number of cigarettes smoked per day and years of smoking experience divided by 20.
Height (cm) | 2 year
  Patient's height measured in centimetres
Weight (kg) | 2 year
  Patient weight measured in kilograms
BMI (kg/m2) | 2 year
  Body mass index is determined using the standard method
Waist circumference (cm) | 2 year
  Waist circumference measured in centimetres using the standard method
Hip circumference (cm) | 2 year
  Hip circumference measured in centimetres using the standard method
Waist circumference to hip circumference ratio (WHR) (number) | 2 year
  Waist circumference to hip circumference index calculated using the standard method
Secondary education (yes/no) | 2 year
  Does the patient have a high school education
Secondary vocational education (yes/no) | 2 year
  Does the patient have a secondary vocational education
Higher education (yes/no) | 2 year
  Does the patient have a university degree
Systolic blood pressure (mmHg) | 2 year
  Systolic blood pressure measured using the standard method
Diastolic blood pressure (mmHg) | 2 year
  Diastolic blood pressure measured using the standard method
Heart rate (number) | 2 year
  Heart rate measured using the standard method
Radial artery pulse (beats per minute). | 2 year
  Radial artery pulse measured using standard methods
Arterial hypertension (yes/no) | 2 year
  History of arterial hypertension
Ultrasound examination of the heart | 2 year
  Ultrasound examination of the heart carried out using standard methods to detect cardiac abnormalities
Total cholesterol (mmol/l) | 2 year
  Total cholesterol measured by standard methods
High-density lipoproteins (HDL) (mmol/l) | 2 year
  High-density lipoproteins measured by standard methods
Low density lipoproteins LDL (mmol/l) | 2 year
  Low density lipoproteins measured by standard methods
Triglycerides (mmol/l) | 2 year
  Triglycerides measured by standard methods
Cholesterol/HDL ratio (number) | 2 year
  Calculated using the standard method
Blood glucose level (mmol/l) | 2 year
  Amount of glucose in the blood measured by the standard method
Glycated haemoglobin (HbA1c), (percent %) | 2 year
  Glycated haemoglobin measured by standard methods
Diabetes mellitus (yes/no) | 2 year
  Indication of diabetes mellitus in the patient's medical history
Taking antihypertensive medication (yes/no) | 2 year
  Indication of antihypertensive medication in the patient's medical history
Taking hypolipidemic medicines (yes/no) | 2 year
  Use of hypolipidemic drugs in a patient's history
Metabolic syndrome (yes/no) | 2 year
  Indicating a history of metabolic syndrome
Presence of post-menopausal diagnosis: arrhythmia or other rhythm disturbances (yes/no) | 2 year
  Post-menopausal diagnosis of arrhythmia or other rhythm disturbances based on medical history
Presence of a post-menopausal diagnosis of coronary heart disease (yes/no) | 2 year
  Presence of post-menopausal diagnosis of coronary heart disease according to medical history
Presence of a post-menopausal diagnosis of myocardial infarction (yes/no) | 2 year
  Post-menopausal diagnosis of myocardial infarction based on medical history
Presence of post-menopausal diagnosis: thromboembolism (yes/no) | 2 year
  Post-menopausal diagnosis of thromboembolism based on medical history
Post-menopausal diagnosis of varicose veins in the lower limbs (yes/no) | 2 year
  Post-menopausal diagnosis of varicose veins in the lower limbs based on medical history
Presence of a post-menopausal diagnosis: Acute cerebral haemorrhage (yes/no) | 2 year
  Post-menopausal diagnosis of acute cerebral haemorrhage on medical history
Deaths from cardiovascular disease in the post-menopausal period (yes/no) | 2 year
  Cardiovascular deaths in the post-menopausal period based on the pathologist's medical history report
A history of cancer (yes/no) | 2 year
  Determined on the basis of the medical history
AGT gene Met235Thr, rs699 polymorphism | 2 year
  Identification of Met235Thr/rs699 polymorphisms in the AGT gene
ACE gene Alu Ins/Del I>D, rs4646994 polymorphism | 2 year
  Identification of Alu Ins/Del I>D, rs4646994 polymorphisms in the ACE gene
NOS3 gene C786T, rs2070744 polymorphism | 2 year
  Identification of C786T, rs2070744 polymorphisms in the NOS3 gene
EDN1 gene Lys198Asn, rs5370 polymorphism | 2 year
  Identification of Lys198Asn, rs5370 polymorphisms in the EDN1 gene
ITGB3 gene Leu33Pro, rs5918 polymorphism | 2 year
  Identification of Leu33Pro, rs5918 polymorphisms in the ITGB3 gene
ITGA2 gene C807T, rs1126643 polymorphism | 2 year
  Identification of C807T, rs1126643 polymorphisms in the ITGA2 gene
FGB gene 455G-A, rs1800790 polymorphism | 2 year
  Identification of 455G-A, rs1800790 polymorphisms in the FGB gene
SERPINE (PAI) 1 gene 675 5G/4G, rs1799768 polymorphism | 2 year
  Identification of 675 5G/4G, rs1799768 polymorphisms in the SERPINE (PAI) 1 gene
CRP gene C3872T, rs1205 polymorphism | 2 year
  Identification of C3872T, rs1205 polymorphisms in the CRP gene
IL17A gene G-197A, rs2275913 polymorphism | 2 year
  Identification of G-197A, rs2275913 polymorphisms in the IL17A gene
IL2 gene T-330G, rs2069762 polymorphism | 2 year
  Identification of T-330G, rs2069762 polymorphisms in the IL2 gene
IL10 gene C-592A, rs1800872 polymorphism | 2 year
  Identification of C-592A, rs1800872 polymorphisms in the IL10 gene
TNF gene G-308A, rs1800629 polymorphism | 2 year
  Identification of G-308A, rs1800629 polymorphisms in the TNF gene
CRP gene A-717G, rs2794521 polymorphism | 2 year
  Identification of A-717G, rs2794521 polymorphisms in the CRP gene
IL6 gene C-174G, rs1800795 polymorphism | 2 year
  Identification of C-174G, rs1800795 polymorphisms in the IL6 gene
TLR2 gene Arg753Gln, rs5743708 polymorphism | 2 year
  Identification of Arg753Gln, rs5743708 polymorphisms in the TLR2 gene
TLR3 gene Phe412Leu, rs3775291 polymorphism | 2 year
  Identification of Phe412Leu, rs3775291 polymorphisms in the TLR3 gene
TLR4 gene Asp299Gly, rs4986790 polymorphism | 2 year
  Identification of Asp299Gly, rs4986790 polymorphisms in the TLR4 gene
TLR6 gene Ser249Pro, rs5743810 polymorphism | 2 year
  Identification of Ser249Pro, rs5743810 polymorphisms in the TLR6 gene
TLR9 gene T-1237C, rs5743836 polymorphism | 2 year
  Identification of T-1237C, rs5743836 polymorphisms in the TLR9 gene

CONTACTS AND LOCATIONS:
Locations (1):
- Sergey Vladimirovich Lopukhov, Ryazan, Ryazan Oblast, Russia

IPD SHARING:
Plan to Share IPD: No